CLINICAL TRIAL: NCT00208273
Title: A Phase II Randomized Study to Compare Skin Late Toxicities of Concomitant Letrozole-Radiotherapy and Radiotherapy Followed by Letrozole as Adjuvant Therapy for Postmenopausal Women With Receptor (ER and/or PgR) Positive Tumors
Brief Title: Concomitant and Sequential Radiohormonotherapy in Adjuvant Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Collaborators: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO-HO-RT/2004/31
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2021-06-02 (Actual); Status verified 2007-12

CONDITIONS: Breast Cancer
Keywords: Postmenopausal breast cancer, radiohormonotherapy sequences; ER+ and/or PgR+,; Postmenopausal Breast cancer,; Adjuvant setting
MeSH Terms: conditions — Breast Neoplasms

ARMS (2):
- A (Experimental): Letrozole 2.5 mg daily for 5 years started three weeks before the first day of adjuvant radiotherapy.
  Interventions: Drug: Letrozole - Concomitant
- B (Experimental): Letrozole 2.5 mg daily for 5 years started three weeks after the last day of adjuvant radiotherapy.
  Interventions: Drug: Letrozole - Sequential

INTERVENTIONS:
Drug: Letrozole - Concomitant
  Arms: A
Drug: Letrozole - Sequential
  Arms: B

SUMMARY:
This trial will compare grade 2 or greater late skin toxicities of concomitant letrozole-radiotherapy and radiotherapy followed by letrozole as adjuvant therapy for postmenopausal women with receptor (estrogen receptor [ER] and/or progesterone receptor [PgR]) positive tumors. Each drug will be prescribed for 5 years.

DETAILED DESCRIPTION:
This trial is an open-label randomized multicenter phase II study.

A ratio of 1 to 1 will be used for the randomization process between the two arms:

* Arm A : Letrozole 2.5 mg daily for 5 years started three weeks before the first day of adjuvant radiotherapy.
* Arm B : Letrozole 2.5 mg daily for 5 years started three weeks after the last day of adjuvant radiotherapy.

All patients will be followed every 3 months for toxicities, disease status and for survival until death.

ELIGIBILITY:
Inclusion Criteria:

* Compliant postmenopausal women
* Conservative breast cancer surgery
* Extension evaluation of disease will be proven negative
* Patients with tumor negative margins
* Patients will be classified as T1, T2, T3; Sentinel node negative, N0, N1 or N2; M0.
* Receptor positive tumors (ER and/or PgR = 10 fmol/mg cytosol protein; or = 10% of the tumor cells positive by immunocytochemical evaluation).
* Adequate marrow function (polynuclear neutrophils >= 1200.10^9/l, platelets >= 100.10^9/l, and hemoglobin >= 10 g/dl).
* Hepatic function (bilirubin >= 30 µmol/l, ALT (SGPT) or AST (SGOT) >= 1.5 x upper limit of the institution) and cholesterol level <2 x upper limit of the institution.
* Must be geographically accessible for follow-up.
* Written and dated informed consent

Exclusion Criteria:

* Patients with distant metastases.
* Bilateral breast cancer (concomitant or prior) except in situ lesion, either ductal or lobular, of the contralateral breast.
* Patients staged T4 or N3 or treated by not conservative surgery (radical mastectomy).
* Patients with neoadjuvant chemotherapy or hormonal therapy.
* Patients with previous or concomitant other (not breast cancer) malignancy within the past 5 years EXCEPT adequately treated basal or squamous cell carcinoma of the skin or in situ carcinoma of the cervix. Patients who have had a previous other malignancy must have been disease free for at least five years.
* Patients with other non-malignant systemic diseases (cardiovascular, renal, hepatic, lung embolism, etc.) which would prevent prolonged follow-up.
* Patients treated with systemic investigational drugs within the past 30 days.
* Breast cancer chemoprevention with anti-estrogens
* Hormone replacement therapy (HRT) not stopped at least 4 weeks before randomization
* Patients known to be HIV positive (no specific tests are required to determine the eligibility).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-01 (Actual); Primary Completion 2007-01 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Sub-cutaneous late toxicity | 2 years

SECONDARY OUTCOMES:
Early toxicity
Lung late toxicity
Cosmetic results
Local failure
Relapse-free survival
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: David AZRIA, MD,PhD, Principal Investigator — CRLC Val d'Aurelle
Locations (1):
- CRLC Val d'Aurelle, Montpellier, France

REFERENCES:
- [Background] Azria D, Pelegrin A, Dubois JB, Mirimanoff RO, Ozsahin M. Radiation therapy and tamoxifen: concurrent or sequential? It's no longer the question! J Clin Oncol. 2005 Jun 20;23(18):4239-41; author reply 4241-2. doi: 10.1200/JCO.2004.00.8623. No abstract available. PMID 15961779
- [Background] Azria D, Larbouret C, Cunat S, Ozsahin M, Gourgou S, Martineau P, Evans DB, Romieu G, Pujol P, Pelegrin A. Letrozole sensitizes breast cancer cells to ionizing radiation. Breast Cancer Res. 2005;7(1):R156-63. doi: 10.1186/bcr969. Epub 2004 Dec 7. PMID 15642164
- [Background] Azria D, Gourgou S, Sozzi WJ, Zouhair A, Mirimanoff RO, Kramar A, Lemanski C, Dubois JB, Romieu G, Pelegrin A, Ozsahin M. Concomitant use of tamoxifen with radiotherapy enhances subcutaneous breast fibrosis in hypersensitive patients. Br J Cancer. 2004 Oct 4;91(7):1251-60. doi: 10.1038/sj.bjc.6602146. PMID 15328527
- [Background] Azria D, Lemanski C, Zouhair A, Gutowski M, Belkacemi Y, Dubois JB, Romieu G, Ozsahin M. [Adjuvant treatment of breast cancer by concomitant hormonotherapy and radiotherapy: state of the art]. Cancer Radiother. 2004 Jun;8(3):188-96. doi: 10.1016/j.canrad.2004.01.003. French. PMID 15217586
- [Derived] Bourgier C, Kerns S, Gourgou S, Lemanski C, Gutowski M, Fenoglietto P, Romieu G, Crompton N, Lacombe J, Pelegrin A, Ozsahin M, Rosenstein B, Azria D. Concurrent or sequential letrozole with adjuvant breast radiotherapy: final results of the CO-HO-RT phase II randomized trial. Ann Oncol. 2016 Mar;27(3):474-80. doi: 10.1093/annonc/mdv602. Epub 2015 Dec 17. PMID 26681684
- [Derived] Azria D, Belkacemi Y, Romieu G, Gourgou S, Gutowski M, Zaman K, Moscardo CL, Lemanski C, Coelho M, Rosenstein B, Fenoglietto P, Crompton NE, Ozsahin M. Concurrent or sequential adjuvant letrozole and radiotherapy after conservative surgery for early-stage breast cancer (CO-HO-RT): a phase 2 randomised trial. Lancet Oncol. 2010 Mar;11(3):258-65. doi: 10.1016/S1470-2045(10)70013-9. Epub 2010 Feb 6. PMID 20138810